CLINICAL TRIAL: NCT02532348
Title: Platelets Study: Influence of the Antiretroviral Treatment on the Platelet Physiology During HIV Infection
Acronym: PLAQUETTE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1108080
Record Dates: First submitted 2015-08-20; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; HIV; antiretroviral therapy; platelets; Immune activation; Inflammatory state
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV Patients with antiretroviral therapy: Blood samples in HIV patients under 2 NRTIs (Nucleosidic analogs of Transcriptase Reverse Inhibitors) and 1 PI or 2 NRTIs and 1 NNRTI, for at least one year with a plasmatic viral load under 40 cp/ml.
  Interventions: Other: Blood samples
- HIV patients without antiretroviral therapy: Blood samples in HIV patients never treated by antiretroviral therapy
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples

SUMMARY:
HIV infection is associated with an immune activation and an inflammatory response - despite an active antiretroviral therapy - which may lead notably but not exclusively to cardiovascular diseases. It has been shown that the use of Protease Inhibitors (PI) instead of Non Nucleosidic Inhibitors (NNRTI) may increase the risk of myocardial infarction. Platelets may play a role in the occurrence of the inflammatory state: they contain big amounts of chemokines, growth factors, and adhesion proteins. Today, the contribution of platelets to the inflammatory state associated with HIV infection has been little studied. Thus, it has been shown that platelets in HIV patients are able to release interleukin (IL)-18. The group has shown with others that the platelet function could be altered during HIV infection. Inversely, it doesn't know how antiretroviral therapy interacts with platelets.

The aim of the study is to evaluate, according to the antiretroviral therapy, the impact on the platelets activation markers.

ELIGIBILITY:
Inclusion Criteria:

* Unchanged antiretroviral therapy for at least one year
* Plasmatic viral load < 40 copies/ml.
* signature of informed consent

Exclusion Criteria:

* Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HVC) coinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study populations:
  * HIV patients under 2 NRTIs (Nucleosidic analogs of Transcriptase Reverse Inhibitors) and 1 PI or 2 NRTIs and 1 NNRTI, for at least one year with a plasmatic viral load under 40 cp/ml.
  * Untreated HIV patients
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Plasmatic level of sCD40L | day 1
  Comparison of plasmatic level of soluble Cluster Differentiation (sCD40L) between 2 groups : HIV patients treated by antiretroviral therapy and HIV patients untreated. sCD40L is measured by enzyme linked immunosorbent assay (ELISA) in ng/ml.

SECONDARY OUTCOMES:
sCD40L level | day 1
  Comparison of plasmatic level of sCD40L between 2 groups : patients treated with 2 Nucleosidic analogs of Transcriptase Reverse Inhibitors (NRTIs ) and 1 Protease Inhibitors (PI) and patients treated with 2 NRTIs and 1 NNRTI. sCD40L is measured by ELISA in ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lucht, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France